CLINICAL TRIAL: NCT01945723
Title: Tissue Characterization From Various Parts of the Gastrointestinal Tract in Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-ZH-553-CTIL
Record Dates: First submitted 2013-09-15; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Endoscopy; Gastrointestinal tract; Bacterial markers; volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Tissue, liquid and stool samples from Gastrointestinal tract.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy volunteers

SUMMARY:
Tissue characterization will be performed, from different regions of the gastrointestinal tract in healthy volunteers.

DETAILED DESCRIPTION:
During an endoscopic examination tissue samples will be taken from different regions of the gastrointestinal mucosa. The tissue samples will be used to characterize bacterial markers in the various intestinal segments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers,
* Age: 20-60 years,
* Consent to perform endoscopic examination.

Exclusion Criteria:

* Antibiotics - a month prior to participation in the study,
* A chronic health condition.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 10 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Bacterial markers in different intestinal segments. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroentherology, Tel Aviv, Israel